CLINICAL TRIAL: NCT06919575
Title: A Individualized Physical Function Improvement Program for Frailty Elderly Using Goal Attainment Scaling (GAS) as Evaluation Method: Protocol for a Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CYYY-Frailty-GAS
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-01

CONDITIONS: Elderly

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the intervention group (Experimental): the intervention group will receive individualized interventions.
  Interventions: Combination Product: Multicomponent frailty intervention
- The control group (No Intervention): The control group will receive routine diagnosis and treatment

INTERVENTIONS:
Combination Product: Multicomponent frailty intervention — First, the underlying causes of the patient's frailty should be analyzed. Individualized goals should be established using Goal Attainment Scaling (GAS), followed by implementation of tailored measures. For patients presenting with malnutrition or mood-related disorders, comprehensive nutritional and psychological assessments must be conducted, with subsequent nutritional support or pharmacological treatment initiated when clinically indicated.
  The patients of the intervention group with poor physical function would receive exercise prescription tailored to the subjects' physical ability from a trained specialist. For Participants requiring exercise-based interventions, a moderate and gradually increasing intensity exercise regimen home-basethree times a week, over a 12-week duration will be administer under telehealth-based monitoring.
  Arms: the intervention group

SUMMARY:
Frailty refers to the age-related decline in physiological functions，that is associated with adverse outcomes. Frailty is a dynamic reversible state, that requires a comprehensive individualized management. Goal Attainment Scaling (GAS) is a structured, individualized method for setting and evaluating progress toward personalized goals.

We conducted a randomized clinical trial of an individualized intervention program using GAS as evaluation method designed to improve physical functional in frailty elderly. A total of 160 individuals aged ≥60 years, who fulfill the Fried scale of frailty will be recruited from Beijing Chaoyang Hospital, Capital Medical University. All participants set personalized goals through GAS. Patients in the intervention group receive individualized interventions, implement tailored measures based on personalized goals to reverse the frailty state.The participants will be followed-up for 3 months and 24 months.

This protocol would be established to examine the efficiency of targeted individualized intervention for frailty based on the GAS. If a positive consequence could be obtained, the results of this study will provide critical data for management of frailty in the elderly, that can be carried out in routine clinical practice.

ELIGIBILITY:
The inclusion criteria were the following: (1)≥60-years old; (2) recognized as frailty by Fried scale.

The exclusion criteria were the following: (1) considered with life expectancy < 1 year such as advanced cancer patients; (2) difficult to communicate with such as patients with severe cognitive impairment (Mini Mental State Examination score ≤ 17); (3) severe hearing disord.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Goal Attainment Scaling (GAS) Formulation of intervention objectives and attainment of goals was assessed using the Goal Attainment Scaling (GAS). GAS is a structured, individualized method for setting and evaluating progress toward personalized goals. | The GAS score was calculated according to a standardized formula and assessed at baseline, 3 months, and 24 months.
  A pool of potential goals was developed by the research team based on the International Classification of Functioning, Disability, and Health (ICF). Each participants selected three goals through collaborative discussions among physicians, the individual, and caregivers. Participants were actively involved in the goal-setting and goal-rating process with the guidance of the research team. Participants also should weigh their goals by importance and difficulty at baseline. Goals were weighted by multiplying the importance level and the anticipated difficulty level, both graded on a 0-3 scale. For each goal, create a 5-point scale(-2 to +2) to describe potential outcomes: -2: Much worse than expected;-1: Somewhat worse than expected; 0: Expected level of success;+1: Somewhat better than expected; +2: Much better than expected. An aggregated T score with a mean of 50 and an SD of 10 was obtained.The extent to which goals are achieved is standardised into a T score by the formula

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kang Y, Qi ZC, Guo MT, Wang XJ. An individualized physical function improvement program for frailty elderly using goal attainment scaling (GAS) as evaluation method: protocol for a randomized controlled trial. BMC Geriatr. 2025 Jul 15;25(1):528. doi: 10.1186/s12877-025-06203-1. PMID 40665225